CLINICAL TRIAL: NCT00021528
Title: Sequenced Treatment Alternatives to Relieve Depression
Brief Title: Sequenced Treatment Alternatives to Relieve Depression (STAR*D)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01MH90003 (NIH); DSIR AT
Record Dates: First submitted 2001-07-20; First posted 2001-07-23 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2006-09

CONDITIONS: Depression
Keywords: Sequential Treatment; Major Depression; Treatment Resistant Depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Citalopram; Buspirone; Lithium; Mirtazapine; Nortriptyline; Sertraline; Tranylcypromine; Cognitive Behavioral Therapy; Triiodothyronine

INTERVENTIONS:
Drug: citalopram
Drug: BuproprionSR
Drug: buspirone
Drug: Lithium
Drug: mirtazapine
Drug: nortriptyline
Drug: sertraline
Drug: tranylcypromine
Drug: VenlafaxineXR
Behavioral: Cognitive Therapy
Drug: T3 (Triiodothyronine)

SUMMARY:
STAR*D focuses on non-psychotic major depressive disorder in adults who are seen in outpatient settings. The primary purpose of this research study is to determine which treatments work best if the first treatment with medication does not produce an acceptable response. Participants will first receive citalopram, an SSRI medication; if symptoms remain after 8-12 weeks of treatment, up to four other levels of treatment will be offered, including cognitive therapy and other medications. There are no placebo treatments. Some patients may require a combination of two or more treatments to obtain full benefit. Participation could last from 15 to 27 months and involve up to 30 clinic visits. Participants will be interviewed by telephone throughout the study about their symptoms, daily functioning, treatment side effects, use of the health care system, and satisfaction with treatment. There will be a one-year follow up for participants once their depression has been successfully treated

DETAILED DESCRIPTION:
The STAR*D project will enroll 4,000 outpatients (ages 18 -75) diagnosed with nonpsychotic Major Depressive Disorder. Participants will be initially treated (open label) with citalopram, the Level 1 treatment, for a minimum of 8 weeks. Patients who experience minimal benefit will be strongly encouraged to complete 12 weeks of treatment in order to maximize the chances of symptom remission (unless no benefit at all is seen after 8 weeks). All participants will also receive a brief depression educational program.

At each level change, participants will be asked to indicate the unacceptability of the potential treatment strategies (e.g, to augment or to switch medications). Participants will then be eligible for random assignment to one of the acceptable and medically safe treatment options.

Level 2: Participants who either did not have an adequate response to or could not tolerate citalopram are eligible for Level 2. The Level 2 treatment strategies are:

i) Medication and Psychotherapy Switch: switch to sertraline, venlafaxineXR, bupropionSR, or cognitive therapy (CT).

ii) Medication and Psychotherapy Augmentation: add to citalopram either a) buspirone, b) bupropionSR, or c) CT.

iii) Medication Only Switch or Medication Only Augmentation options are available for participants for whom CT is unacceptable.

iv)Psychotherapy Only Switch or Psychotherapy Only Augmentation options are available for participants for whom additional medication is unacceptable at this point in the study (participants must be willing to continue citalopram)

Level 2A: Participants without a satisfactory response to their Level 2 treatment are eligible for random assignment to additional treatment at Level 2A (if medically safe and acceptable). Level 2A is included so that all participants entering Level 3 have had an opportunity to respond to at least 2 medications. Level 2A consists of Medication Switch to one of two antidepressant medications (venlafaxineXR or bupropion SR).

Level 3: Participants without satisfactory response to Level 2 and,if appropriate Level 2A, are eligible for random assignment to one of the following treatments (if acceptable and medically safe):

i) Medication Switch to: a) mirtazapine or b) nortriptyline, a tricyclic antidepressant.

ii) Medication Augmentation: Add (to current Level 2 or Level 2A medication) either: a) lithium or b) thyroid hormone (T3).

Level 4: Participants without an adequate response to Level 3 are eligible for random assignment to Level 4 treatment (if acceptable and medically safe). Level 4 includes two Medication Switch options: to tranylcypromine [a monoamine oxidase inhibitor (MAOI)], or to mirtazapine plus venlafaxineXR.

After Level 4, participants without an adequate response will discuss other acceptable treatment options with their physician.

Once an adequate response is achieved at Levels 2, 2A, 3 or 4, participants are eligible to enter the 12-month follow-up, during which time they will remain on their current treatment(s) and will be asked about their symptoms and other relevant information monthly by telephone. ONLY PATIENTS BEING TREATED AT THE PARTICIPATING CLINICS ARE ELIGIBLE FOR THIS STUDY.

ELIGIBILITY:
- Outpatients aged 18 to 75 years old with nonpsychotic major depressive disorder (HAMD score 14 or greater)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000
Dates: Start 2001-07; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: A. John Rush, MD, Study Director — University of Texas Southwestern Medical Center Department of Psychiatry
Locations (41):
- United States (41):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - Tuscaloosa VA Mental Health Clinic - Veterans Only, Tuscaloosa, Alabama
  - Tuscaloosa VA Primary Care Center, Tuscaloosa, Alabama
  - Psychiatric Centers at San Diego, Chula Vista, California
  - Harbor UCLA Family Health Care Center, Harbor City, California
  - UCLA General Outpatient Psychiatry Clinic, Los Angeles, California
  - UCLA Internal Medicine Clinic, Los Angeles, California
  - UCSD Outpatient Psychiatric Services, San Diego, California
  - Veterans Affairs Medical Center/FIRM Primary Care Clinic, San Diego, California
  - Harbor UCLA Medical Center, Torrance, California
  - Northwestern Outpatient Treatment Care Center, Chicago, Illinois
  - University of Illinois at Chicago Clinic, Chicago, Illinois
  - Evanston Outpatient Clinic, Evanston, Illinois
  - COMCARE of Sedgwick County, Wichita, Kansas
  - Psychiatric Outpatient Clinic, Wichita, Kansas
  - Swampscott Family Doctors, Boston, Massachusetts
  - Internal Medicine Associates, Boston, Massachusetts
  - MGH/Charlestown Clinic, Charlestown, Massachusetts
  - MGH/Salem Professional, Salem, Massachusetts
  - General Psychiatric Ambulatory Clinic, Ann Arbor, Michigan
  - Briarwood Family Practice Clinic, Ann Arbor, Michigan
  - LIJ/Zucker Hillside Adult Ambulatory Care Center, Glen Oaks, New York
  - LIJ North Shore Medical Group, Lake Success, New York
  - UNC Chapel Hill General Medicine Clinic, Chapel Hill, North Carolina
  - UNC Chapel Hill Adult Diagnostic & Treatment Clinic, Chapel Hill, North Carolina
  - UNC Chapel Hill Family Practice Clinic, Chapel Hill, North Carolina
  - Springer Family Medicine, Tulsa, Oklahoma
  - Laureate Psychiatric Clinic & Hospital, Tulsa, Oklahoma
  - Warren Clinic, Tulsa, Oklahoma
  - Diversified Human Services Clinic, Pittsburgh, Pennsylvania
  - Latterman Family Health Center, Pittsburgh, Pennsylvania
  - Bellefield Clinic of WPIC, Pittsburgh, Pennsylvania
  - AMPN Corkery, Heise & Dainesi, Upper Saint Clair, Pennsylvania
  - Psychiatric Consultants, P.C., Nashville, Tennessee
  - Vanderbilt University Medical Center-Mental Health Center, Nashville, Tennessee
  - Vine Hill Community Clinic, Nashville, Tennessee
  - Centerstone/Luton Mental Health Services, Nashville, Tennessee
  - The Holiner Psychiatric Group, Dallas, Texas
  - UT Southwestern Family Medicine Clinic, Dallas, Texas
  - MCV Primary Care Clinic, Richmond, Virginia
  - MCV Family Counseling, Richmond, Virginia

REFERENCES:
- [Background] Adli M, Rush AJ, Moller HJ, Bauer M. Algorithms for optimizing the treatment of depression: making the right decision at the right time. Pharmacopsychiatry. 2003 Nov;36 Suppl 3:S222-9. doi: 10.1055/s-2003-45134. PMID 14677083
- [Background] Fava M, Rush AJ, Trivedi MH, Nierenberg AA, Thase ME, Sackeim HA, Quitkin FM, Wisniewski S, Lavori PW, Rosenbaum JF, Kupfer DJ. Background and rationale for the sequenced treatment alternatives to relieve depression (STAR*D) study. Psychiatr Clin North Am. 2003 Jun;26(2):457-94, x. doi: 10.1016/s0193-953x(02)00107-7. PMID 12778843
- [Background] Rush AJ, Trivedi M, Fava M. Depression, IV: STAR*D treatment trial for depression. Am J Psychiatry. 2003 Feb;160(2):237. doi: 10.1176/appi.ajp.160.2.237. No abstract available. PMID 12562566
- [Background] Lavori PW, Rush AJ, Wisniewski SR, Alpert J, Fava M, Kupfer DJ, Nierenberg A, Quitkin FM, Sackeim HA, Thase ME, Trivedi M. Strengthening clinical effectiveness trials: equipoise-stratified randomization. Biol Psychiatry. 2001 Nov 15;50(10):792-801. doi: 10.1016/s0006-3223(01)01223-9. PMID 11720698
- [Background] Rush AJ, Fava M, Wisniewski SR, Lavori PW, Trivedi MH, Sackeim HA, Thase ME, Nierenberg AA, Quitkin FM, Kashner TM, Kupfer DJ, Rosenbaum JF, Alpert J, Stewart JW, McGrath PJ, Biggs MM, Shores-Wilson K, Lebowitz BD, Ritz L, Niederehe G; STAR*D Investigators Group. Sequenced treatment alternatives to relieve depression (STAR*D): rationale and design. Control Clin Trials. 2004 Feb;25(1):119-42. doi: 10.1016/s0197-2456(03)00112-0. PMID 15061154
- [Background] Wisniewski SR, Stegman D, Trivedi M, Husain MM, Eng H, Shores-Wilson K, Luther J, Biggs MM, Burroughs D, Ritz AL, Fava M, Quitkin F, Rush AJ; STAR*D Investigators. Methods of testing feasibility for sequenced treatment alternatives to relieve depression (STAR*D). J Psychiatr Res. 2004 May-Jun;38(3):241-8. doi: 10.1016/j.jpsychires.2003.06.001. PMID 15003429
- [Background] Wisniewski SR, Eng H, Meloro L, Gatt R, Ritz L, Stegman D, Trivedi M, Biggs MM, Friedman E, Shores-Wilson K, Warden D, Bartolowits D, Martin JP, Rush AJ. Web-based communications and management of a multi-center clinical trial: the Sequenced Treatment Alternatives to Relieve Depression (STAR*D) project. Clin Trials. 2004;1(4):387-98. doi: 10.1191/1740774504cn035oa. PMID 16279277
- [Background] Nierenberg AA, Trivedi MH, Ritz L, Burroughs D, Greist J, Sackeim H, Kornstein S, Schwartz T, Stegman D, Fava M, Wisniewski SR. Suicide risk management for the sequenced treatment alternatives to relieve depression study: applied NIMH guidelines. J Psychiatr Res. 2004 Nov-Dec;38(6):583-9. doi: 10.1016/j.jpsychires.2004.03.004. PMID 15458854
- [Background] Yates WR, Mitchell J, Rush AJ, Trivedi MH, Wisniewski SR, Warden D, Hauger RB, Fava M, Gaynes BN, Husain MM, Bryan C. Clinical features of depressed outpatients with and without co-occurring general medical conditions in STAR*D. Gen Hosp Psychiatry. 2004 Nov-Dec;26(6):421-9. doi: 10.1016/j.genhosppsych.2004.06.008. PMID 15567207
- [Background] Fava M, Alpert JE, Carmin CN, Wisniewski SR, Trivedi MH, Biggs MM, Shores-Wilson K, Morgan D, Schwartz T, Balasubramani GK, Rush AJ. Clinical correlates and symptom patterns of anxious depression among patients with major depressive disorder in STAR*D. Psychol Med. 2004 Oct;34(7):1299-308. doi: 10.1017/s0033291704002612. PMID 15697056
- [Background] Friedman EF, Thase ME, Biggs MM, Carmin C, Hollon SD, Kornblith SJ, Petersen T, Veenstra G, Wisniewski SR, and Rush AJ. The implementation of cognitive therapy in STAR*D. Cognitive Therapy and Research, 28:819-833, 2004.
- [Background] Zisook S, Rush AJ, Albala A, Alpert J, Balasubramani GK, Fava M, Husain M, Sackeim H, Trivedi M, Wisniewski S. Factors that differentiate early vs. later onset of major depression disorder. Psychiatry Res. 2004 Dec 15;129(2):127-40. doi: 10.1016/j.psychres.2004.07.004. PMID 15590040
- [Background] Davis LL, Rush JA, Wisniewski SR, Rice K, Cassano P, Jewell ME, Biggs MM, Shores-Wilson K, Balasubramani GK, Husain MM, Quitkin FM, McGrath PJ. Substance use disorder comorbidity in major depressive disorder: an exploratory analysis of the Sequenced Treatment Alternatives to Relieve Depression cohort. Compr Psychiatry. 2005 Mar-Apr;46(2):81-9. doi: 10.1016/j.comppsych.2004.07.025. PMID 15723023
- [Background] Perlis RH, Fraguas R, Fava M, Trivedi MH, Luther JF, Wisniewski SR, Rush AJ. Prevalence and clinical correlates of irritability in major depressive disorder: a preliminary report from the Sequenced Treatment Alternatives to Relieve Depression study. J Clin Psychiatry. 2005 Feb;66(2):159-66; quiz 147, 273-4. PMID 15705000
- [Background] Warden D, Rush AJ, Trivedi M, Ritz L, Stegman D, Wisniewski SR. Quality improvement methods as applied to a multicenter effectiveness trial--STAR*D. Contemp Clin Trials. 2005 Feb;26(1):95-112. doi: 10.1016/j.cct.2004.11.011. Epub 2005 Jan 27. PMID 15837455
- [Background] Gaynes BN, Rush AJ, Trivedi M, Wisniewski SR, Balasubramani GK, Spencer DC, Petersen T, Klinkman M, Warden D, Schneider RK, Castro DB, Golden RN. A direct comparison of presenting characteristics of depressed outpatients from primary vs. specialty care settings: preliminary findings from the STAR*D clinical trial. Gen Hosp Psychiatry. 2005 Mar-Apr;27(2):87-96. doi: 10.1016/j.genhosppsych.2004.10.003. PMID 15763119
- [Background] Kornstein SG, Harvey AT, Rush AJ, Wisniewski SR, Trivedi MH, Svikis DS, McKenzie ND, Bryan C, Harley R. Self-reported premenstrual exacerbation of depressive symptoms in patients seeking treatment for major depression. Psychol Med. 2005 May;35(5):683-92. doi: 10.1017/s0033291704004106. PMID 15918345
- [Background] Rush AJ, Zimmerman M, Wisniewski SR, Fava M, Hollon SD, Warden D, Biggs MM, Shores-Wilson K, Shelton RC, Luther JF, Thomas B, Trivedi MH. Comorbid psychiatric disorders in depressed outpatients: demographic and clinical features. J Affect Disord. 2005 Jul;87(1):43-55. doi: 10.1016/j.jad.2005.03.005. PMID 15894381
- [Background] Marcus SM, Young EA, Kerber KB, Kornstein S, Farabaugh AH, Mitchell J, Wisniewski SR, Balasubramani GK, Trivedi MH, Rush AJ. Gender differences in depression: findings from the STAR*D study. J Affect Disord. 2005 Aug;87(2-3):141-50. doi: 10.1016/j.jad.2004.09.008. PMID 15982748
- [Background] Lesser IM, Leuchter AF, Trivedi MH, Davis LL, Wisniewski SR, Balasubramani GK, Petersen T, Stegman D, Rush AJ. Characteristics of insured and noninsured outpatients with depression in STAR(*)D. Psychiatr Serv. 2005 Aug;56(8):995-1004. doi: 10.1176/appi.ps.56.8.995. PMID 16088018
- [Background] Novick JS, Stewart JW, Wisniewski SR, Cook IA, Manev R, Nierenberg AA, Rosenbaum JF, Shores-Wilson K, Balasubramani GK, Biggs MM, Zisook S, Rush AJ; STAR*D investigators. Clinical and demographic features of atypical depression in outpatients with major depressive disorder: preliminary findings from STAR*D. J Clin Psychiatry. 2005 Aug;66(8):1002-11. doi: 10.4088/jcp.v66n0807. PMID 16086615
- [Background] Husain MM, Rush AJ, Sackeim HA, Wisniewski SR, McClintock SM, Craven N, Holiner J, Mitchell JR, Balasubramani GK, Hauger R. Age-related characteristics of depression: a preliminary STAR*D report. Am J Geriatr Psychiatry. 2005 Oct;13(10):852-60. doi: 10.1176/appi.ajgp.13.10.852. PMID 16223963
- [Background] Gaynes, B.N., Davis, L., Rush A.J., Trivedi, M., Fava, M., Wisniewski, S.R. The aims and design of the Sequenced Treatment Alternatives to Relieve Depression (STAR*D) study. Primary Psychiatry, 12(2):36-41, 2005.
- [Background] Friedman EF, Thase ME, Biggs MM, Carmin C, Hollon SD, Kornblith SJ, Petersen T, Veenstra G, Wisniewski SR, Rush AJ. The implementation of cognitive therapy in STAR*D. Cognit Ther Res 2004;28:819-33.
- [Background] Gaynes BN, Davis L, Rush AJ, Trivedi MH, Fava M, Wisniewski SR. The aims and design of the Sequenced Treatment Alternatives to Relieve Depression (STAR*D) study. Primary Psychiatry 2005;12(2):36-41. http://www.primarypsychiatry.com/pdf/art_4845.pdf
- [Background] Gilmer WS, Trivedi MH, Rush AJ, Wisniewski SR, Luther J, Howland RH, Yohanna D, Khan A, Alpert J. Factors associated with chronic depressive episodes: a preliminary report from the STAR-D project. Acta Psychiatr Scand. 2005 Dec;112(6):425-33. doi: 10.1111/j.1600-0447.2005.00633.x. PMID 16279871
- [Background] Hollon SD, Shelton RC, Wisniewski S, Warden D, Biggs MM, Friedman ES, Husain M, Kupfer DJ, Nierenberg AA, Petersen TJ, Shores-Wilson K, Rush AJ. Presenting characteristics of depressed outpatients as a function of recurrence: preliminary findings from the STAR*D clinical trial. J Psychiatr Res. 2006 Feb;40(1):59-69. doi: 10.1016/j.jpsychires.2005.07.008. Epub 2005 Oct 21. PMID 16243357
- [Background] Rush AJ, Bernstein IH, Trivedi MH, Carmody TJ, Wisniewski S, Mundt JC, Shores-Wilson K, Biggs MM, Woo A, Nierenberg AA, Fava M. An evaluation of the quick inventory of depressive symptomatology and the hamilton rating scale for depression: a sequenced treatment alternatives to relieve depression trial report. Biol Psychiatry. 2006 Mar 15;59(6):493-501. doi: 10.1016/j.biopsych.2005.08.022. Epub 2005 Sep 30. PMID 16199008
- [Background] Davis LL, Frazier E, Husain MM, Warden D, Trivedi M, Fava M, Cassano P, McGrath PJ, Balasubramani GK, Wisniewski SR, Rush AJ. Substance use disorder comorbidity in major depressive disorder: a confirmatory analysis of the STAR*D cohort. Am J Addict. 2006 Jul-Aug;15(4):278-85. doi: 10.1080/10550490600754317. PMID 16867922
- [Result] Trivedi MH, Rush AJ, Wisniewski SR, Nierenberg AA, Warden D, Ritz L, Norquist G, Howland RH, Lebowitz B, McGrath PJ, Shores-Wilson K, Biggs MM, Balasubramani GK, Fava M; STAR*D Study Team. Evaluation of outcomes with citalopram for depression using measurement-based care in STAR*D: implications for clinical practice. Am J Psychiatry. 2006 Jan;163(1):28-40. doi: 10.1176/appi.ajp.163.1.28. PMID 16390886
- [Result] Pilowsky DJ, Wickramaratne PJ, Rush AJ, Hughes CW, Garber J, Malloy E, King CA, Cerda G, Sood AB, Alpert JE, Wisniewski SR, Trivedi MH, Talati A, Carlson MM, Liu HH, Fava M, Weissman MM. Children of currently depressed mothers: a STAR*D ancillary study. J Clin Psychiatry. 2006 Jan;67(1):126-36. doi: 10.4088/jcp.v67n0119. PMID 16426099
- [Result] Trivedi MH, Rush AJ, Wisniewski SR, Warden D, McKinney W, Downing M, Berman SR, Farabaugh A, Luther JF, Nierenberg AA, Callan JA, Sackeim HA. Factors associated with health-related quality of life among outpatients with major depressive disorder: a STAR*D report. J Clin Psychiatry. 2006 Feb;67(2):185-95. doi: 10.4088/jcp.v67n0203. PMID 16566612
- [Result] Rush AJ, Trivedi MH, Wisniewski SR, Stewart JW, Nierenberg AA, Thase ME, Ritz L, Biggs MM, Warden D, Luther JF, Shores-Wilson K, Niederehe G, Fava M; STAR*D Study Team. Bupropion-SR, sertraline, or venlafaxine-XR after failure of SSRIs for depression. N Engl J Med. 2006 Mar 23;354(12):1231-42. doi: 10.1056/NEJMoa052963. PMID 16554525
- [Result] Weissman MM, Pilowsky DJ, Wickramaratne PJ, Talati A, Wisniewski SR, Fava M, Hughes CW, Garber J, Malloy E, King CA, Cerda G, Sood AB, Alpert JE, Trivedi MH, Rush AJ; STAR*D-Child Team. Remissions in maternal depression and child psychopathology: a STAR*D-child report. JAMA. 2006 Mar 22;295(12):1389-98. doi: 10.1001/jama.295.12.1389. PMID 16551710
- [Result] Trivedi MH, Fava M, Wisniewski SR, Thase ME, Quitkin F, Warden D, Ritz L, Nierenberg AA, Lebowitz BD, Biggs MM, Luther JF, Shores-Wilson K, Rush AJ; STAR*D Study Team. Medication augmentation after the failure of SSRIs for depression. N Engl J Med. 2006 Mar 23;354(12):1243-52. doi: 10.1056/NEJMoa052964. PMID 16554526
- [Result] Fava M, Rush AJ, Wisniewski SR, Nierenberg AA, Alpert JE, McGrath PJ, Thase ME, Warden D, Biggs M, Luther JF, Niederehe G, Ritz L, Trivedi MH. A comparison of mirtazapine and nortriptyline following two consecutive failed medication treatments for depressed outpatients: a STAR*D report. Am J Psychiatry. 2006 Jul;163(7):1161-72. doi: 10.1176/ajp.2006.163.7.1161. PMID 16816220
- [Result] McGrath PJ, Stewart JW, Fava M, Trivedi MH, Wisniewski SR, Nierenberg AA, Thase ME, Davis L, Biggs MM, Shores-Wilson K, Luther JF, Niederehe G, Warden D, Rush AJ. Tranylcypromine versus venlafaxine plus mirtazapine following three failed antidepressant medication trials for depression: a STAR*D report. Am J Psychiatry. 2006 Sep;163(9):1531-41; quiz 1666. doi: 10.1176/ajp.2006.163.9.1531. PMID 16946177
- [Result] Nierenberg AA, Fava M, Trivedi MH, Wisniewski SR, Thase ME, McGrath PJ, Alpert JE, Warden D, Luther JF, Niederehe G, Lebowitz B, Shores-Wilson K, Rush AJ. A comparison of lithium and T(3) augmentation following two failed medication treatments for depression: a STAR*D report. Am J Psychiatry. 2006 Sep;163(9):1519-30; quiz 1665. doi: 10.1176/ajp.2006.163.9.1519. PMID 16946176
- [Result] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Result] McMahon FJ, Buervenich S, Charney D, Lipsky R, Rush AJ, Wilson AF, Sorant AJM, Papanicolaou GJ, Laje G, Fava M, Trivedi MH, Wisniewski SR, Manji H. Variation in the gene encoding the serotonin 2A receptor is associated with outcome of antidepressant treatment. Am J Hum Genet. 2006 May;78(5):804-814. doi: 10.1086/503820. Epub 2006 Mar 20. PMID 16642436
- [Result] Alpert JE, Biggs MM, Davis L, Shores-Wilson K, Harlan WR, Schneider GW, Ford AL, Farabaugh A, Stegman D, Ritz AL, Husain MM, Macleod L, Wisniewski SR, Rush AJ; STAR*D Investigators. Enrolling research subjects from clinical practice: ethical and procedural issues in the Sequenced Treatment Alternatives to Relieve Depression (STAR*D) trial. Psychiatry Res. 2006 Feb 28;141(2):193-200. doi: 10.1016/j.psychres.2005.04.007. Epub 2006 Feb 2. PMID 16457894
- [Result] Khan AY, Carrithers J, Preskorn SH, Lear R, Wisniewski SR, John Rush A, Stegman D, Kelley C, Kreiner K, Nierenberg AA, Fava M. Clinical and demographic factors associated with DSM-IV melancholic depression. Ann Clin Psychiatry. 2006 Apr-Jun;18(2):91-8. doi: 10.1080/10401230600614496. PMID 16754414
- [Result] Wisniewski SR, Leon AC, Otto MW, Trivedi MH. Prevention of missing data in clinical research studies. Biol Psychiatry. 2006 Jun 1;59(11):997-1000. doi: 10.1016/j.biopsych.2006.01.017. Epub 2006 Mar 29. PMID 16566901
- [Result] Fava M, Rush AJ. Current status of augmentation and combination treatments for major depressive disorder: a literature review and a proposal for a novel approach to improve practice. Psychother Psychosom. 2006;75(3):139-53. doi: 10.1159/000091771. PMID 16636629
- [Result] Nierenberg AA, Trivedi MH, Fava M, Biggs MM, Shores-Wilson K, Wisniewski SR, Balasubramani GK, Rush AJ. Family history of mood disorder and characteristics of major depressive disorder: a STAR*D (sequenced treatment alternatives to relieve depression) study. J Psychiatr Res. 2007 Apr-Jun;41(3-4):214-21. doi: 10.1016/j.jpsychires.2006.02.005. Epub 2006 May 11. PMID 16690084
- [Result] Claassen CA, Trivedi MH, Rush AJ, Husain MM, Zisook S, Young E, Leuchter A, Wisniewski SR, Balasubramani GK, Alpert J. Clinical differences among depressed patients with and without a history of suicide attempts: findings from the STAR*D trial. J Affect Disord. 2007 Jan;97(1-3):77-84. doi: 10.1016/j.jad.2006.05.026. Epub 2006 Jul 7. PMID 16824617
- [Result] Gilmer WS, Kemp DE. STAR*D: What Have We Learned Thus Far? International Drug Therapy Newsletter 41:75-82, 2006.
- [Result] Fava M, Rush AJ, Alpert JE, Carmin CN, Balasubramani GK, Wisniewski SR, Trivedi MH, Biggs MM, Shores-Wilson K. What clinical and symptom features and comorbid disorders characterize outpatients with anxious major depressive disorder: a replication and extension. Can J Psychiatry. 2006 Nov;51(13):823-35. doi: 10.1177/070674370605101304. PMID 17195602
- [Result] Murphy SA, Oslin DW, Rush AJ, Zhu J; MCATS. Methodological challenges in constructing effective treatment sequences for chronic psychiatric disorders. Neuropsychopharmacology. 2007 Feb;32(2):257-62. doi: 10.1038/sj.npp.1301241. Epub 2006 Nov 8. PMID 17091129
- [Result] Zisook S, Rush AJ, Lesser I, Wisniewski SR, Trivedi M, Husain MM, Balasubramani GK, Alpert JE, Fava M. Preadult onset vs. adult onset of major depressive disorder: a replication study. Acta Psychiatr Scand. 2007 Mar;115(3):196-205. doi: 10.1111/j.1600-0447.2006.00868.x. PMID 17302619
- [Derived] Phaterpekar T, Nunez JJ, Morton E, Liu YS, Cao B, Frey BN, Milev RV, Muller DJ, Rotzinger S, Soares CN, Taylor VH, Uher R, Kennedy SH, Lam RW. Machine Learning Prediction of Quality of Life Improvement During Antidepressant Treatment of Patients With Major Depressive Disorder: A STAR*D and CAN-BIND-1 Report. J Clin Psychiatry. 2023 Nov 15;85(1):23m14864. doi: 10.4088/JCP.23m14864. PMID 37967350
- [Derived] Shah SB, Peddada TN, Song C, Mensah M, Sung H, Yavi M, Yuan P, Zarate CA Jr, Mickey BJ, Burmeister M, Akula N, McMahon FJ. Exome-wide association study of treatment-resistant depression suggests novel treatment targets. Sci Rep. 2023 Aug 1;13(1):12467. doi: 10.1038/s41598-023-38984-z. PMID 37528149
- [Derived] Salem H, Huynh T, Topolski N, Mwangi B, Trivedi MH, Soares JC, Rush AJ, Selvaraj S. Temporal multi-step predictive modeling of remission in major depressive disorder using early stage treatment data; STAR*D based machine learning approach. J Affect Disord. 2023 Mar 1;324:286-293. doi: 10.1016/j.jad.2022.12.076. Epub 2022 Dec 28. PMID 36584711
- [Derived] Oliva V, Fanelli G, Kasper S, Zohar J, Souery D, Montgomery S, Albani D, Forloni G, Ferentinos P, Rujescu D, Mendlewicz J, Kas MJ, De Ronchi D, Fabbri C, Serretti A. Social withdrawal as a trans-diagnostic predictor of short-term remission: a meta-analysis of five clinical cohorts. Int Clin Psychopharmacol. 2022 Mar 1;37(2):38-45. doi: 10.1097/YIC.0000000000000384. PMID 34855649
- [Derived] Fanelli G, Domschke K, Minelli A, Gennarelli M, Martini P, Bortolomasi M, Maron E, Squassina A, Kasper S, Zohar J, Souery D, Montgomery S, Albani D, Forloni G, Ferentinos P, Rujescu D, Mendlewicz J, De Ronchi D, Baune BT; European College of Neuropsychopharmacology (ECNP) Pharmacogenomics & Transcriptomics Thematic Working Group; Serretti A, Fabbri C. A meta-analysis of polygenic risk scores for mood disorders, neuroticism, and schizophrenia in antidepressant response. Eur Neuropsychopharmacol. 2022 Feb;55:86-95. doi: 10.1016/j.euroneuro.2021.11.005. Epub 2021 Nov 26. PMID 34844152
- [Derived] Kappelmann N, Czamara D, Rost N, Moser S, Schmoll V, Trastulla L, Stochl J, Lucae S; CHARGE inflammation working group; Binder EB, Khandaker GM, Arloth J. Polygenic risk for immuno-metabolic markers and specific depressive symptoms: A multi-sample network analysis study. Brain Behav Immun. 2021 Jul;95:256-268. doi: 10.1016/j.bbi.2021.03.024. Epub 2021 Mar 29. PMID 33794315
- [Derived] Rush AJ, South C, Jha MK, Jain SB, Trivedi MH. What to Expect When Switching to a Second Antidepressant Medication Following an Ineffective Initial SSRI: A Report From the Randomized Clinical STAR*D Study. J Clin Psychiatry. 2020 Aug 11;81(5):19m12949. doi: 10.4088/JCP.19m12949. PMID 32780949
- [Derived] Porcelli S, Kasper S, Zohar J, Souery D, Montgomery S, Ferentinos P, Rujescu D, Mendlewicz J, Merlo Pich E, Pollentier S, Penninx BWJH, Serretti A. Social dysfunction in mood disorders and schizophrenia: Clinical modulators in four independent samples. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Apr 20;99:109835. doi: 10.1016/j.pnpbp.2019.109835. Epub 2019 Dec 11. PMID 31836507
- [Derived] Baez LM, Heller AS. Impact of age at onset on the phenomenology of depression in treatment-seeking adults in the STAR*D trial. J Affect Disord. 2020 Feb 1;262:381-388. doi: 10.1016/j.jad.2019.10.036. Epub 2019 Oct 26. PMID 31740109
- [Derived] Mason BL, Davidov A, Minhajuddin A, Trivedi MH. Focusing on insomnia symptoms to better understand depression: A STAR*D report. J Affect Disord. 2020 Jan 1;260:183-186. doi: 10.1016/j.jad.2019.08.094. Epub 2019 Aug 30. PMID 31499373
- [Derived] Wallace MP, Moodie EEM, Stephens DA. Model selection for G-estimation of dynamic treatment regimes. Biometrics. 2019 Dec;75(4):1205-1215. doi: 10.1111/biom.13104. Epub 2019 Sep 12. PMID 31222720
- [Derived] Callan JA, Kazantzis N, Park SY, Moore CG, Thase ME, Minhajuddin A, Kornblith S, Siegle GJ. A Propensity Score Analysis of Homework Adherence-Outcome Relations in Cognitive Behavioral Therapy for Depression. Behav Ther. 2019 Mar;50(2):285-299. doi: 10.1016/j.beth.2018.05.010. Epub 2018 Jun 5. PMID 30824246
- [Derived] Fabbri C, Kasper S, Kautzky A, Bartova L, Dold M, Zohar J, Souery D, Montgomery S, Albani D, Raimondi I, Dikeos D, Rujescu D, Uher R, Lewis CM, Mendlewicz J, Serretti A. Genome-wide association study of treatment-resistance in depression and meta-analysis of three independent samples. Br J Psychiatry. 2019 Jan;214(1):36-41. doi: 10.1192/bjp.2018.256. Epub 2018 Nov 23. PMID 30468137
- [Derived] Fabbri C, Tansey KE, Perlis RH, Hauser J, Henigsberg N, Maier W, Mors O, Placentino A, Rietschel M, Souery D, Breen G, Curtis C, Lee SH, Newhouse S, Patel H, O'Donovan M, Lewis G, Jenkins G, Weinshilboum RM, Farmer A, Aitchison KJ, Craig I, McGuffin P, Schruers K, Biernacka JM, Uher R, Lewis CM. Effect of cytochrome CYP2C19 metabolizing activity on antidepressant response and side effects: Meta-analysis of data from genome-wide association studies. Eur Neuropsychopharmacol. 2018 Aug;28(8):945-954. doi: 10.1016/j.euroneuro.2018.05.009. Epub 2018 Jun 28. PMID 30135031
- [Derived] Nie Z, Vairavan S, Narayan VA, Ye J, Li QS. Predictive modeling of treatment resistant depression using data from STAR*D and an independent clinical study. PLoS One. 2018 Jun 7;13(6):e0197268. doi: 10.1371/journal.pone.0197268. eCollection 2018. PMID 29879133
- [Derived] Fabbri C, Tansey KE, Perlis RH, Hauser J, Henigsberg N, Maier W, Mors O, Placentino A, Rietschel M, Souery D, Breen G, Curtis C, Sang-Hyuk L, Newhouse S, Patel H, Guipponi M, Perroud N, Bondolfi G, O'Donovan M, Lewis G, Biernacka JM, Weinshilboum RM, Farmer A, Aitchison KJ, Craig I, McGuffin P, Uher R, Lewis CM. New insights into the pharmacogenomics of antidepressant response from the GENDEP and STAR*D studies: rare variant analysis and high-density imputation. Pharmacogenomics J. 2018 May 22;18(3):413-421. doi: 10.1038/tpj.2017.44. Epub 2017 Nov 21. PMID 29160301
- [Derived] Steiner AJ, Recacho J, Vanle B, Dang J, Wright SM, Miller JS, Kauzor K, Reid M, Bashmi LE, Mirocha J, Danovitch I, IsHak WW. Quality of Life, Functioning, and Depressive Symptom Severity in Older Adults With Major Depressive Disorder Treated With Citalopram in the STAR*D Study. J Clin Psychiatry. 2017 Jul;78(7):897-903. doi: 10.4088/JCP.16m11335. PMID 28858443
- [Derived] Lopez E, Steiner AJ, Manier K, Shapiro BB, Vanle B, Parisi T, Dang J, Chang T, Ganjian S, Mirocha J, Danovitch I, IsHak WW. Quality of life and functioning of Hispanic patients with Major Depressive Disorder before and after treatment. J Affect Disord. 2018 Jan 1;225:117-122. doi: 10.1016/j.jad.2017.08.031. Epub 2017 Aug 14. PMID 28826087
- [Derived] Garcia-Gonzalez J, Tansey KE, Hauser J, Henigsberg N, Maier W, Mors O, Placentino A, Rietschel M, Souery D, Zagar T, Czerski PM, Jerman B, Buttenschon HN, Schulze TG, Zobel A, Farmer A, Aitchison KJ, Craig I, McGuffin P, Giupponi M, Perroud N, Bondolfi G, Evans D, O'Donovan M, Peters TJ, Wendland JR, Lewis G, Kapur S, Perlis R, Arolt V, Domschke K; Major Depressive Disorder Working Group of the Psychiatric Genomic Consortium; Breen G, Curtis C, Sang-Hyuk L, Kan C, Newhouse S, Patel H, Baune BT, Uher R, Lewis CM, Fabbri C. Pharmacogenetics of antidepressant response: A polygenic approach. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Apr 3;75:128-134. doi: 10.1016/j.pnpbp.2017.01.011. Epub 2017 Jan 31. PMID 28159590
- [Derived] IsHak WW, Bonifay W, Collison K, Reid M, Youssef H, Parisi T, Cohen RM, Cai L. The recovery index: A novel approach to measuring recovery and predicting remission in major depressive disorder. J Affect Disord. 2017 Jan 15;208:369-374. doi: 10.1016/j.jad.2016.08.081. Epub 2016 Oct 15. PMID 27810720
- [Derived] Danovitch I, Steiner AJ, Kazdan A, Goldenberg M, Haglund M, Mirocha J, Collison K, Vanle B, Dang J, IsHak WW. Analysis of Patient-reported Outcomes of Quality of Life and Functioning Before and After Treatment of Major Depressive Disorder Comorbid With Alcohol Use Disorders. J Addict Med. 2017 Jan/Feb;11(1):47-54. doi: 10.1097/ADM.0000000000000268. PMID 27763941
- [Derived] Coughlin CG, Jakubovski E, Bloch MH. Time Course and Predictors of Suicidal Ideation During Citalopram Treatment in the STAR*D Trial. J Clin Psychiatry. 2016 Oct;77(10):e1262-e1269. doi: 10.4088/JCP.15m10075. PMID 27631142
- [Derived] Diaz FJ. Measuring the individual benefit of a medical or behavioral treatment using generalized linear mixed-effects models. Stat Med. 2016 Oct 15;35(23):4077-92. doi: 10.1002/sim.7005. Epub 2016 Jun 20. PMID 27323698
- [Derived] Olbert CM, Rasmussen A, Gala GJ, Tupler LA. Treatment outcome variation between depression symptom combinations in the STAR*D study. J Affect Disord. 2016 Sep 1;201:1-7. doi: 10.1016/j.jad.2016.04.050. Epub 2016 Apr 26. PMID 27155023
- [Derived] Pearson R, Palmer RH, Brick LA, McGeary JE, Knopik VS, Beevers CG. Additive genetic contribution to symptom dimensions in major depressive disorder. J Abnorm Psychol. 2016 May;125(4):495-501. doi: 10.1037/abn0000161. PMID 27124715
- [Derived] Cocchi E, Fabbri C, Han C, Lee SJ, Patkar AA, Masand PS, Pae CU, Serretti A. Genome-wide association study of antidepressant response: involvement of the inorganic cation transmembrane transporter activity pathway. BMC Psychiatry. 2016 Apr 18;16:106. doi: 10.1186/s12888-016-0813-x. PMID 27091189
- [Derived] Fervaha G, Foussias G, Takeuchi H, Agid O, Remington G. Motivational deficits in major depressive disorder: Cross-sectional and longitudinal relationships with functional impairment and subjective well-being. Compr Psychiatry. 2016 Apr;66:31-8. doi: 10.1016/j.comppsych.2015.12.004. Epub 2015 Dec 18. PMID 26995233
- [Derived] Fried EI, van Borkulo CD, Epskamp S, Schoevers RA, Tuerlinckx F, Borsboom D. Measuring depression over time . . . Or not? Lack of unidimensionality and longitudinal measurement invariance in four common rating scales of depression. Psychol Assess. 2016 Nov;28(11):1354-1367. doi: 10.1037/pas0000275. Epub 2016 Jan 28. PMID 26821198
- [Derived] Chekroud AM, Zotti RJ, Shehzad Z, Gueorguieva R, Johnson MK, Trivedi MH, Cannon TD, Krystal JH, Corlett PR. Cross-trial prediction of treatment outcome in depression: a machine learning approach. Lancet Psychiatry. 2016 Mar;3(3):243-50. doi: 10.1016/S2215-0366(15)00471-X. Epub 2016 Jan 21. PMID 26803397
- [Derived] Ulbricht CM, Dumenci L, Rothschild AJ, Lapane KL. Changes in depression subtypes for women during treatment with citalopram: a latent transition analysis. Arch Womens Ment Health. 2016 Oct;19(5):769-78. doi: 10.1007/s00737-016-0606-8. Epub 2016 Jan 22. PMID 26802021
- [Derived] Xu MY, Umbach DM, Murphy E, McMahon F, Shugart YY. A Novel Mixture Model to Estimate the Time to Drug Effect Onset and Its Association with Covariates. Hum Hered. 2015;80(2):90-9. doi: 10.1159/000440880. Epub 2016 Jan 16. PMID 26771572
- [Derived] Baer L, Trivedi MH, Huz I, Rush AJ, Wisniewski SR, Fava M. Prevalence and impact of obsessive-compulsive symptoms in depression: a STAR*D report. J Clin Psychiatry. 2015 Dec;76(12):1668-74. doi: 10.4088/JCP.14m09670. PMID 26717526
- [Derived] Minelli A, Magri C, Barbon A, Bonvicini C, Segala M, Congiu C, Bignotti S, Milanesi E, Trabucchi L, Cattane N, Bortolomasi M, Gennarelli M. Proteasome system dysregulation and treatment resistance mechanisms in major depressive disorder. Transl Psychiatry. 2015 Dec 1;5(12):e687. doi: 10.1038/tp.2015.180. PMID 26624926
- [Derived] Fried EI, Epskamp S, Nesse RM, Tuerlinckx F, Borsboom D. What are 'good' depression symptoms? Comparing the centrality of DSM and non-DSM symptoms of depression in a network analysis. J Affect Disord. 2016 Jan 1;189:314-20. doi: 10.1016/j.jad.2015.09.005. Epub 2015 Oct 1. PMID 26458184
- [Derived] Ulbricht CM, Rothschild AJ, Lapane KL. The association between latent depression subtypes and remission after treatment with citalopram: A latent class analysis with distal outcome. J Affect Disord. 2015 Dec 1;188:270-7. doi: 10.1016/j.jad.2015.08.039. Epub 2015 Sep 1. PMID 26384013
- [Derived] Boles RG, Zaki EA, Kerr JR, Das K, Biswas S, Gardner A. Increased prevalence of two mitochondrial DNA polymorphisms in functional disease: Are we describing different parts of an energy-depleted elephant? Mitochondrion. 2015 Jul;23:1-6. doi: 10.1016/j.mito.2015.04.005. Epub 2015 Apr 29. PMID 25934187
- [Derived] Fabbri C, Crisafulli C, Gurwitz D, Stingl J, Calati R, Albani D, Forloni G, Calabro M, Martines R, Kasper S, Zohar J, Juven-Wetzler A, Souery D, Montgomery S, Mendlewicz J, Girolamo GD, Serretti A. Neuronal cell adhesion genes and antidepressant response in three independent samples. Pharmacogenomics J. 2015 Dec;15(6):538-48. doi: 10.1038/tpj.2015.15. Epub 2015 Apr 7. PMID 25850031
- [Derived] Congiu C, Minelli A, Bonvicini C, Bortolomasi M, Sartori R, Maj C, Scassellati C, Maina G, Trabucchi L, Segala M, Gennarelli M. The role of the potassium channel gene KCNK2 in major depressive disorder. Psychiatry Res. 2015 Feb 28;225(3):489-92. doi: 10.1016/j.psychres.2014.11.061. Epub 2014 Dec 9. PMID 25535009
- [Derived] Fried EI, Nesse RM. Depression is not a consistent syndrome: An investigation of unique symptom patterns in the STAR*D study. J Affect Disord. 2015 Feb 1;172:96-102. doi: 10.1016/j.jad.2014.10.010. Epub 2014 Oct 14. PMID 25451401
- [Derived] Arias B, Fabbri C, Serretti A, Drago A, Mitjans M, Gasto C, Catalan R, Fananas L. DISC1-TSNAX and DAOA genes in major depression and citalopram efficacy. J Affect Disord. 2014 Oct;168:91-7. doi: 10.1016/j.jad.2014.06.048. Epub 2014 Jul 5. PMID 25043320
- [Derived] Drago A, Cocchi E, Crisafulli C, Serretti A. A molecular pathway analysis of the glutamatergic-monoaminergic interplay serves to investigate the number of depressive records during citalopram treatment. J Neural Transm (Vienna). 2015 Mar;122(3):465-75. doi: 10.1007/s00702-014-1267-2. Epub 2014 Jul 2. PMID 24986638
- [Derived] IsHak WW, Mirocha J, James D, Tobia G, Vilhauer J, Fakhry H, Pi S, Hanson E, Nashawati R, Peselow ED, Cohen RM. Quality of life in major depressive disorder before/after multiple steps of treatment and one-year follow-up. Acta Psychiatr Scand. 2015 Jan;131(1):51-60. doi: 10.1111/acps.12301. Epub 2014 Jun 23. PMID 24954156
- [Derived] Ferguson M, Dennehy EB, Marangell LB, Martinez J, Wisniewski SR. Impact of fatigue on outcome of selective serotonin reuptake inhibitor treatment: secondary analysis of STAR*D. Curr Med Res Opin. 2014 Oct;30(10):2109-18. doi: 10.1185/03007995.2014.936553. Epub 2014 Jul 4. PMID 24949937
- [Derived] Jakubovski E, Bloch MH. Prognostic subgroups for citalopram response in the STAR*D trial. J Clin Psychiatry. 2014 Jul;75(7):738-47. doi: 10.4088/JCP.13m08727. PMID 24912106
- [Derived] Ostergaard SD, Bech P, Trivedi MH, Wisniewski SR, Rush AJ, Fava M. Brief, unidimensional melancholia rating scales are highly sensitive to the effect of citalopram and may have biological validity: implications for the research domain criteria (RDoC). J Affect Disord. 2014 Jul;163:18-24. doi: 10.1016/j.jad.2014.03.049. Epub 2014 Apr 3. PMID 24836083
- [Derived] Tada M, Uchida H, Suzuki T, Abe T, Pollock BG, Mimura M. Baseline difference between patients' and clinicians' rated illness severity scores and subsequent outcomes in major depressive disorder: analysis of the sequenced treatment alternatives to relieve depression data. J Clin Psychopharmacol. 2014 Jun;34(3):297-302. doi: 10.1097/JCP.0000000000000112. No abstract available. PMID 24743720
- [Derived] Fabbri C, Marsano A, Albani D, Chierchia A, Calati R, Drago A, Crisafulli C, Calabro M, Kasper S, Lanzenberger R, Zohar J, Juven-Wetzler A, Souery D, Montgomery S, Mendlewicz J, Serretti A. PPP3CC gene: a putative modulator of antidepressant response through the B-cell receptor signaling pathway. Pharmacogenomics J. 2014 Oct;14(5):463-72. doi: 10.1038/tpj.2014.15. Epub 2014 Apr 8. PMID 24709691
- [Derived] Fried EI, Nesse RM. The impact of individual depressive symptoms on impairment of psychosocial functioning. PLoS One. 2014 Feb 28;9(2):e90311. doi: 10.1371/journal.pone.0090311. eCollection 2014. PMID 24587318
- [Derived] Sakurai H, Uchida H, Abe T, Nakajima S, Suzuki T, Pollock BG, Sato Y, Mimura M. Trajectories of individual symptoms in remitters versus non-remitters with depression. J Affect Disord. 2013 Nov;151(2):506-513. doi: 10.1016/j.jad.2013.06.035. Epub 2013 Jul 22. PMID 23886402
- [Derived] IsHak WW, Mirocha J, Christensen S, Wu F, Kwock R, Behjat J, Pi S, Akopyan A, Peselow ED, Cohen RM, Elashoff D. Patient-reported outcomes of quality of life, functioning, and depressive symptom severity in major depressive disorder comorbid with panic disorder before and after SSRI treatment in the star*d trial. Depress Anxiety. 2014 Aug;31(8):707-16. doi: 10.1002/da.22152. Epub 2013 Jul 16. PMID 23861180
- [Derived] Murphy E, Hou L, Maher BS, Woldehawariat G, Kassem L, Akula N, Laje G, McMahon FJ. Race, genetic ancestry and response to antidepressant treatment for major depression. Neuropsychopharmacology. 2013 Dec;38(13):2598-606. doi: 10.1038/npp.2013.166. Epub 2013 Jul 5. PMID 23827886
- [Derived] Fabbri C, Marsano A, Balestri M, De Ronchi D, Serretti A. Clinical features and drug induced side effects in early versus late antidepressant responders. J Psychiatr Res. 2013 Oct;47(10):1309-18. doi: 10.1016/j.jpsychires.2013.05.020. Epub 2013 Jun 22. PMID 23800418
- [Derived] Ishak WW, Greenberg JM, Cohen RM. Predicting relapse in major depressive disorder using patient-reported outcomes of depressive symptom severity, functioning, and quality of life in the Individual Burden of Illness Index for Depression (IBI-D). J Affect Disord. 2013 Oct;151(1):59-65. doi: 10.1016/j.jad.2013.05.048. Epub 2013 Jun 19. PMID 23790554
- [Derived] Niitsu T, Fabbri C, Bentini F, Serretti A. Pharmacogenetics in major depression: a comprehensive meta-analysis. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Aug 1;45:183-94. doi: 10.1016/j.pnpbp.2013.05.011. Epub 2013 Jun 1. PMID 23733030
- [Derived] Ishak WW, Christensen S, Sayer G, Ha K, Li N, Miller J, Nguyen JM, Cohen RM. Sexual satisfaction and quality of life in major depressive disorder before and after treatment with citalopram in the STAR*D study. J Clin Psychiatry. 2013 Mar;74(3):256-61. doi: 10.4088/JCP.12m07933. PMID 23561231
- [Derived] Trivedi MH, Morris DW, Wisniewski SR, Lesser I, Nierenberg AA, Daly E, Kurian BT, Gaynes BN, Balasubramani GK, Rush AJ. Increase in work productivity of depressed individuals with improvement in depressive symptom severity. Am J Psychiatry. 2013 Jun;170(6):633-41. doi: 10.1176/appi.ajp.2012.12020250. PMID 23558394
- [Derived] Haley CL, Sung SC, Rush AJ, Trivedi MH, Wisniewski SR, Luther JF, Kornstein SG. The clinical relevance of self-reported premenstrual worsening of depressive symptoms in the management of depressed outpatients: a STAR*D report. J Womens Health (Larchmt). 2013 Mar;22(3):219-29. doi: 10.1089/jwh.2011.3186. PMID 23480315
- [Derived] Trivedi MH, Morris DW, Wisniewski SR, Nierenberg AA, Gaynes BN, Kurian BT, Warden D, Stegman D, Shores-Wilson K, Rush AJ. Clinical and sociodemographic characteristics associated with suicidal ideation in depressed outpatients. Can J Psychiatry. 2013 Feb;58(2):113-22. doi: 10.1177/070674371305800209. PMID 23442899
- [Derived] Perlis RH. A clinical risk stratification tool for predicting treatment resistance in major depressive disorder. Biol Psychiatry. 2013 Jul 1;74(1):7-14. doi: 10.1016/j.biopsych.2012.12.007. Epub 2013 Feb 4. PMID 23380715
- [Derived] Cohen RM, Greenberg JM, IsHak WW. Incorporating multidimensional patient-reported outcomes of symptom severity, functioning, and quality of life in the Individual Burden of Illness Index for Depression to measure treatment impact and recovery in MDD. JAMA Psychiatry. 2013 Mar;70(3):343-50. doi: 10.1001/jamapsychiatry.2013.286. PMID 23303512
- [Derived] Smith RM, Papp AC, Webb A, Ruble CL, Munsie LM, Nisenbaum LK, Kleinman JE, Lipska BK, Sadee W. Multiple regulatory variants modulate expression of 5-hydroxytryptamine 2A receptors in human cortex. Biol Psychiatry. 2013 Mar 15;73(6):546-54. doi: 10.1016/j.biopsych.2012.09.028. Epub 2012 Nov 13. PMID 23158458
- [Derived] Uher R, Perlis RH, Placentino A, Dernovsek MZ, Henigsberg N, Mors O, Maier W, McGuffin P, Farmer A. Self-report and clinician-rated measures of depression severity: can one replace the other? Depress Anxiety. 2012 Dec;29(12):1043-9. doi: 10.1002/da.21993. Epub 2012 Aug 29. PMID 22933451
- [Derived] Fabbri C, Drago A, Serretti A. Early antidepressant efficacy modulation by glutamatergic gene variants in the STAR*D. Eur Neuropsychopharmacol. 2013 Jul;23(7):612-21. doi: 10.1016/j.euroneuro.2012.07.006. Epub 2012 Aug 11. PMID 22884879
- [Derived] McClintock SM, Husain MM, Bernstein IH, Wisniewski SR, Trivedi MH, Morris D, Alpert J, Warden D, Luther JF, Kornstein SG, Biggs MM, Fava M, Rush AJ. Assessing anxious features in depressed outpatients. Int J Methods Psychiatr Res. 2011 Dec;20(4):e69-82. doi: 10.1002/mpr.353. Epub 2011 Nov 4. PMID 22057975
- [Derived] Rush AJ, Wisniewski SR, Zisook S, Fava M, Sung SC, Haley CL, Chan HN, Gilmer WS, Warden D, Nierenberg AA, Balasubramani GK, Gaynes BN, Trivedi MH, Hollon SD. Is prior course of illness relevant to acute or longer-term outcomes in depressed out-patients? A STAR*D report. Psychol Med. 2012 Jun;42(6):1131-49. doi: 10.1017/S0033291711002170. Epub 2011 Oct 19. PMID 22008447
- [Derived] Denninger JW, van Nieuwenhuizen AO, Wisniewski SR, Luther JF, Trivedi MH, Rush AJ, Gollan JK, Pizzagalli DA, Fava M. Changes in depressive symptoms and social functioning in the sequenced treatment alternatives to relieve depression study. J Nerv Ment Dis. 2011 Oct;199(10):807-10. doi: 10.1097/NMD.0b013e31822fcbe2. PMID 21964277
- [Derived] Uher R, Perlis RH, Henigsberg N, Zobel A, Rietschel M, Mors O, Hauser J, Dernovsek MZ, Souery D, Bajs M, Maier W, Aitchison KJ, Farmer A, McGuffin P. Depression symptom dimensions as predictors of antidepressant treatment outcome: replicable evidence for interest-activity symptoms. Psychol Med. 2012 May;42(5):967-80. doi: 10.1017/S0033291711001905. Epub 2011 Sep 20. PMID 21929846
- [Derived] Warner-Schmidt JL, Vanover KE, Chen EY, Marshall JJ, Greengard P. Antidepressant effects of selective serotonin reuptake inhibitors (SSRIs) are attenuated by antiinflammatory drugs in mice and humans. Proc Natl Acad Sci U S A. 2011 May 31;108(22):9262-7. doi: 10.1073/pnas.1104836108. Epub 2011 Apr 25. PMID 21518864
- [Derived] Silverstein B, Patel P. Poor response to antidepressant medication of patients with depression accompanied by somatic symptomatology in the STAR*D Study. Psychiatry Res. 2011 May 15;187(1-2):121-4. doi: 10.1016/j.psychres.2010.12.026. Epub 2011 Jan 8. PMID 21216475
- [Derived] Kuk AY, Li J, Rush AJ. Recursive subsetting to identify patients in the STAR*D: a method to enhance the accuracy of early prediction of treatment outcome and to inform personalized care. J Clin Psychiatry. 2010 Nov;71(11):1502-8. doi: 10.4088/JCP.10m06168blu. PMID 21114950
- [Derived] Garriock HA, Tanowitz M, Kraft JB, Dang VC, Peters EJ, Jenkins GD, Reinalda MS, McGrath PJ, von Zastrow M, Slager SL, Hamilton SP. Association of mu-opioid receptor variants and response to citalopram treatment in major depressive disorder. Am J Psychiatry. 2010 May;167(5):565-73. doi: 10.1176/appi.ajp.2009.08081167. Epub 2010 Mar 1. PMID 20194481
- [Derived] Bergemann ER, Boles RG. Maternal inheritance in recurrent early-onset depression. Psychiatr Genet. 2010 Feb;20(1):31-4. doi: 10.1097/YPG.0b013e3283351153. PMID 20010317
- [Derived] Davis LL, Wisniewski SR, Howland RH, Trivedi MH, Husain MM, Fava M, McGrath PJ, Balasubramani GK, Warden D, Rush AJ. Does comorbid substance use disorder impair recovery from major depression with SSRI treatment? An analysis of the STAR*D level one treatment outcomes. Drug Alcohol Depend. 2010 Mar 1;107(2-3):161-70. doi: 10.1016/j.drugalcdep.2009.10.003. Epub 2009 Nov 28. PMID 19945804
- [Derived] Leuchter AF, Husain MM, Cook IA, Trivedi MH, Wisniewski SR, Gilmer WS, Luther JF, Fava M, Rush AJ. Painful physical symptoms and treatment outcome in major depressive disorder: a STAR*D (Sequenced Treatment Alternatives to Relieve Depression) report. Psychol Med. 2010 Feb;40(2):239-51. doi: 10.1017/S0033291709006035. Epub 2009 Jun 3. PMID 19493369
- [Derived] Nierenberg AA, Husain MM, Trivedi MH, Fava M, Warden D, Wisniewski SR, Miyahara S, Rush AJ. Residual symptoms after remission of major depressive disorder with citalopram and risk of relapse: a STAR*D report. Psychol Med. 2010 Jan;40(1):41-50. doi: 10.1017/S0033291709006011. Epub 2009 May 22. PMID 19460188
- [Derived] Stewart JW, McGrath PJ, Fava M, Wisniewski SR, Zisook S, Cook I, Nierenberg AA, Trivedi MH, Balasubramani GK, Warden D, Lesser I, John Rush A. Do atypical features affect outcome in depressed outpatients treated with citalopram? Int J Neuropsychopharmacol. 2010 Feb;13(1):15-30. doi: 10.1017/S1461145709000182. Epub 2009 Apr 3. PMID 19341509
- [Derived] Wisniewski SR, Rush AJ, Nierenberg AA, Gaynes BN, Warden D, Luther JF, McGrath PJ, Lavori PW, Thase ME, Fava M, Trivedi MH. Can phase III trial results of antidepressant medications be generalized to clinical practice? A STAR*D report. Am J Psychiatry. 2009 May;166(5):599-607. doi: 10.1176/appi.ajp.2008.08071027. Epub 2009 Apr 1. PMID 19339358
- [Derived] Husain MM, Rush AJ, Wisniewski SR, McClintock SM, Fava M, Nierenberg AA, Davis L, Balasubramani GK, Young E, Albala AA, Trivedi MH. Family history of depression and therapeutic outcome: findings from STAR*D. J Clin Psychiatry. 2009 Feb;70(2):185-95. doi: 10.4088/jcp.07m03571. Epub 2008 Dec 2. PMID 19192454
- [Derived] McGrath PJ, Khan AY, Trivedi MH, Stewart JW, Morris DW, Wisniewski SR, Miyahara S, Nierenberg AA, Fava M, Rush AJ. Response to a selective serotonin reuptake inhibitor (citalopram) in major depressive disorder with melancholic features: a STAR*D report. J Clin Psychiatry. 2008 Dec;69(12):1847-55. doi: 10.4088/jcp.v69n1201. Epub 2008 Nov 18. PMID 19026268
- [Derived] Gilmer WS, Gollan JK, Wisniewski SR, Howland RH, Trivedi MH, Miyahara S, Fleck J, Thase ME, Alpert JE, Nierenberg AA, Warden D, Fava M, Rush AJ. Does the duration of index episode affect the treatment outcome of major depressive disorder? A STAR*D report. J Clin Psychiatry. 2008 Aug;69(8):1246-56. doi: 10.4088/jcp.v69n0807. PMID 18681756
- [Derived] Rush AJ, Wisniewski SR, Warden D, Luther JF, Davis LL, Fava M, Nierenberg AA, Trivedi MH. Selecting among second-step antidepressant medication monotherapies: predictive value of clinical, demographic, or first-step treatment features. Arch Gen Psychiatry. 2008 Aug;65(8):870-80. doi: 10.1001/archpsyc.65.8.870. PMID 18678792
- [Derived] Davis LL, Frazier EC, Gaynes BN, Trivedi MH, Wisniewski SR, Fava M, Barkin J, Kashner TM, Shelton RC, Alpert JE, Rush AJ. Are depressed outpatients with and without a family history of substance use disorder different? A baseline analysis of the STAR*D cohort. J Clin Psychiatry. 2007 Dec;68(12):1931-8. doi: 10.4088/jcp.v68n1214. PMID 18162025
- See also: More information on depression — http://www.nimh.nih.gov/health/topics/depression/index.shtml